The WELL Study (Wellness Education for Liver Health Study): Reducing liver disease in genetically predisposed adults

NCT #05010070

Document date: 07/01/2022

# UNIVERSITY OF MICHIGAN CONSENT TO BE PART OF A RESEARCH STUDY

### 1. KEY INFORMATION ABOUT THE RESEARCHERS AND THIS STUDY

**Study title:** The WELL Study (Wellness Education for Liver Health Study): Reducing liver disease in genetically predisposed adults

Company or agency sponsoring the study: This research is sponsored by a pilot/feasibility study from the Michigan Nutrition Obesity Research Center and by a small research grant (R03) from the National Institutes of Health (NIH).

Names, degrees, and affiliations of the principal investigator and study coordinator (if applicable): Principal Investigator: Laura Saslow, Ph.D., Assistant Professor in the Department of Health Behavior and Biological Sciences in the School of Nursing, University of Michigan, Ann Arbor

# 1.1 Key Study Information

You may be eligible to take part in a research study. This form contains important information that will help you decide whether to join the study. Take the time to carefully review this information. You should talk to the researchers about the study and ask them any questions you have. You may also wish to talk to others such as your family, friends, or other doctors about joining this study. If you decide to join the study, you will be asked to sign this form before you can start study-related activities. Before you do, be sure you understand what the research study is about.

A research study is different from the regular medical care you receive from your doctor. Research studies hope to make discoveries and learn new information about diseases and how to treat them. You should consider the reasons why you might want to join a research study or why it is not the best decision for you at this time.

Research studies do not always offer the possibility of treating your disease or condition. Research studies also have different kinds of risks and risk levels, depending on the type of the study. You may also need to think about other requirements for being in the study. For example, some studies require you to travel to scheduled visits at the study site in Ann Arbor or elsewhere. This may require you to arrange travel, change work schedules, find child care, or make other plans. In your decision to participate in this study, consider all of these matters carefully.

This research is studying whether changing an individual's behaviors may have an impact as a treatment for Non-alcoholic Fatty Liver Disease (NAFLD). This research will test whether following a very low-carbohydrate diet for 4 months helps patients with NAFLD control their condition, lose weight, and/or improves quality of life. Your health-related information, including questionnaire responses, blood samples, and MRI results, will be collected for this research study.

There can be risks associated with joining any research study. The type of risk may impact whether you decide to join the study. For this study, some of these risks may include side effects such as cramping, headaches, or bad breath, inconvenience due to at-home tasks and travel for appointments, or loss of privacy. More detailed information will be provided later in this document.

IRBMED Informed Consent Template—3-9-2018

Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

This study may offer some benefit to you now or others in the future by improving your health outcomes and/or providing information that will affect how physicians treat NAFLD in the future. More information will be provided later in this document.

We expect the amount of time you will participate in the study will be about six months – approximately one month to determine if you are eligible, four months as part of the study, and one month for your follow up appointments.

You can decide not to be in this study. Alternatives to joining this study include continuing care for your non-alcoholic fatty liver disease as normal.

Even if you decide to join the study now, you are free to leave at any time if you change your mind.

More information about this study continues in Section 2 of this document.

### 2. PURPOSE OF THIS STUDY

**2.1 Study purpose:** Non-alcoholic fatty liver disease (NAFLD) affects, on average, 30% of the population. Some will go on to get advanced liver disease whereas others will not. We are studying the effects of genetics and environment on burden of NAFLD, specifically how modifying diet can affect the disease. We will investigate how a very low carbohydrate diet can interact with your genome to improve your liver health. Your genome is all of your hereditary information, encoded in DNA. This study will support participants in following a diet and lifestyle program.

# 3. WHO MAY PARTICIPATE IN THE STUDY

Taking part in this study is completely **voluntary**. You do not have to participate if you don't want to. You may also leave the study at any time. If you leave the study before it is finished, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

### 3.1 Who can take part in this study?

You were contacted about this study because you are in the Michigan Genomics Initiative (MGI) database. Additionally, you have been identified as a potential subject from completing the prescreening survey that verified you are at least 18 years of age or older, with elevated liver function tests, fluent in the English language, have regular access to the internet, and have no physical limitations that might interfere with your participation in the study.

You may not participate in the study if you are pregnant, have type 1 diabetes, heart failure or cancer.

# 3.2 How many people are expected to take part in this study?

We expect up to 40 people to take part in this study.

# 4. INFORMATION ABOUT STUDY PARTICIPATION

# 4.1 What will happen to me in this study?

You have already completed several tasks as part of your eligibility screening for this trial. Next, you'll review and sign this consent form with the study coordinator over the phone (you'll sign this form online) and make two appointments with us.

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

- Your first appointment will be a virtual visit with one of the study doctors. Your medical
  history and health will be evaluated. We'll check for high blood pressure, cardiovascular
  disease (angina, myocardial infarction, stroke, heart failure), and other conditions which
  may be causing elevated liver function tests.
- After your first appointment, you will get fasting blood tests done- about 7 teaspoons of blood will be drawn. These tests can be done at one of any Michigan Medicine blood draw clinics that's most convenient for you (<a href="https://mlabs.umich.edu/blood-draw-station">https://mlabs.umich.edu/blood-draw-station</a>). You'll need to fast for 8 hours before these tests (you can only have water during these 8 hours) and complete them within one week of your virtual visit. The blood tests will help us (1) evaluate the cause of your elevated liver functions (2) test for diabetes and (3) test for elevated cholesterol. We will draw about 4 tsp of blood for these tests.
  - We will draw extra blood at these appointments, about 2 additional tsp. Some of this blood will be tested for an appetite-suppressing hormone.
  - Other blood will be drawn to make "induced pluripotent stem cells" or iPS cells and will be used to determine if your cells develop disease or respond to treatments the way you do. To create iPS cells from your blood after it has been draw, certain genes are introduced into the blood to "reprogram" these cells to become pluripotent, that is, able to become any cell in the body, such as brain, liver, or heart cells. Animal testing is conducted to verify that the "reprogramed" cells are pluripotent. The iPS cell research is an optional component of this trial. You may still participate in the WELL study if you decide not to have excess blood drawn for iPS cell research.
    - If you choose to participate in this optional research, then you'll need to make an appointment to get your blood drawn at the Taubman Center in Michigan Medicine's main hospital. These will take place on the morning of a weekday within the week or two after your virtual visit. A member of our staff may meet you at your blood draw to collect your iPS cell sample.

You may be diagnosed with a condition that is not non-alcoholic fatty liver disease. This will make you ineligible.

After your virtual visit and fasting blood tests:

- We'll send you a short survey to ask for your contact information and the name of your physician. The study team will get permission from your primary care provider for you to participate in the trial.
- You will complete either two 24-hour dietary recalls OR you'll track your food for three days on the MyFitnessPal website. We will let you know which step you'll be completing. If you complete the dietary recalls, a member of our team will reach out to you twice over the phone to discuss everything you ate the day before. If you complete the dietary tracking, you'll set up an account on MyFitnessPal (we'll send you directions) and track everything you eat for three days. You'll create and share a pin number with us so that we can view your tracking logs without logging into your account. Here's MyFitnessPal's privacy statement: <a href="https://www.myfitnesspal.com/privacy-policy">https://www.myfitnesspal.com/privacy-policy</a>
- If you are a woman of childbearing potential, we'll send you an at-home urine pregnancy test. This test will be for you to complete the morning of your second appointment. We'll

ask you to send a photo of the result to our study email address (<a href="mailto:info\_well@nutritionstudy.org">info\_well@nutritionstudy.org</a>). You will not be able to proceed to your MRI appointment and won't be eligible to join the study if your pregnancy screening is positive.

- If no other cause of elevated liver function tests is found during your first appointment and blood tests, except for NAFLD, you will come to the hospital for your second appointment, where you will receive a liver MRI, which is the current gold standard for non-invasive measurement of liver steatosis (fatty liver), fibrosis and cirrhosis (liver scarring). The MRI appointment will take up to two hours, but usually lasts less than an hour.
  - You will need to fast for at least 4 hours prior to your MRI (including avoiding water).
  - The MRI team will go over the procedure with you and will ask you questions about your health history. You may be unable to receive the MRI as a result of your health history and will not be eligible to join the trial.
  - If you are ineligible to join the trial based on your MRI results or your MRI screening, we will send you a \$20 Amazon gift card as a thank you for your efforts.

Your eligibility for the study will be determined based on the evaluation of your MRI results. If you are eligible to join the study, we'll mail you a digital scale. This scale automatically sends us the weights you take. After you step on the scale and we receive your weight, you'll be ready to begin the online diet and lifestyle program.

### **Study Procedures**

By being in the program, you will receive care at our NAFLD liver clinic; we will provide state-of-the-art care and resources about NAFLD to all participants.

You will receive the standard patient packet as a part of your virtual appointment, which includes:

- 1) NAFLD disease information including diagnosis, clinical manifestations, natural history, and treatments;
- 2) NAFLD physical activity recommendations including walking programs and physical activity logs;
- 3) Weight tracking logs; and
- 4) Resources for diet and exercise programs

We will send you several items in the mail at the start of the study, including a cookbook, ketostix (to measure ketone levels, which will help you track yourself on a very low carbohydrate diet), and a bodyweight scale.

You will receive your first class email on a Sunday, which will introduce you to the diet and lifestyle program and help you transition to a very low-carbohydrate diet. In this program, you'll be encouraged to eat foods like non-starchy vegetables, leafy greens, cheese, meats, berries, nuts, and seeds and to avoid starchy foods like pasta, bread, rice, etc. Cutting out carbs in your diet can bring you into "ketosis," which means your body will start burning fat for energy instead of carbohydrates.

You will receive a class email every Sunday for 16 weeks, with articles to read, videos to watch, a skill to practice, and a survey to check in with us. You will also have contact with a diet coach over email, who will be available to answer your questions and provide support.

If you're taking blood-glucose lowering medications other than metformin, we'll send you a glucometer at the beginning of the study, so that you can keep track of your blood glucose throughout. We'll ask that you check your blood glucose while you're fasted and postprandial (2 hours after eating) a few times a week. Each week, in the check-in survey, we'll ask you to tell us your highest and lowest blood glucose readings from the past week (both fasted numbers and postprandial numbers). We'll keep an eye on your blood glucose reports and reach out if any medication adjustments are necessary or if we recommend speaking with your primary care provider.

At the end of the 4-month program, we will ask you to repeat many of the measure you completed at the start of the trial, including the virtual visit, liver MRI (and urine pregnancy test), fasting blood tests (about 2.5 tsp for standard tests and an additional 2 tsp for iPS cell testing), online survey, and tracking your diet for 3 days with MyFitnessPal or 24-hour dietary recalls. As a reminder, MyFitnessPal is a free website that allows you to track the food that you eat and share your food logs with the study team. Additionally, the online survey will ask questions about your satisfaction with and feedback about the study and program. If you elect to participate in the iPS cell research, your 4-month blood draw will also take place at the hospital during a weekday. Otherwise, you can attend whichever clinic is most convenient for you.

You may be asked if you'd like to participate in an optional exit interview. This interview will be about your experience in the program and should take less than 30 minutes. The interview will be recorded, though only the study team or professional transcribers will hear your interview. This is entirely optional and you will be able to opt out at any time.

# How will your study supplies be provided to you?

Some of your study materials and emails may be sent directly to you through vendors such as:

- Amazon (for mailing gift certificates and cookbooks)
  - Amazon privacy policy: <a href="https://www.amazon.com/gp/help/customer/display.html?nodeld=GX7NJQ4ZB8M">https://www.amazon.com/gp/help/customer/display.html?nodeld=GX7NJQ4ZB8M</a>
     <a href="https://www.amazon.com/gp/help/customer/display.html?nodeld=GX7NJQ4ZB8M">https://www.amazon.com/gp/help/customer/display.html?nodeld=GX7NJQ4ZB8M</a>
- BodyTrace (body weight scale)
  - BodyTrace has signed a non-disclosure agreement with the University of Michigan, visible here: <a href="https://www.dropbox.com/s/zsam9epdjxjgzgy/NDA%20UM-Body%20Trace%205500020633Fully%20Executed%20033021.pdf?dl=0">https://www.dropbox.com/s/zsam9epdjxjgzgy/NDA%20UM-Body%20Trace%205500020633Fully%20Executed%20033021.pdf?dl=0</a>
- GSuite/Gmail and Postmarkapp (for emails),
  - Google privacy policy: https://policies.google.com/privacy?hl=en-US
  - Postmarkapp privacy policy: <a href="https://wildbit.com/privacy-policy">https://wildbit.com/privacy-policy</a>
- Qualtrics (for surveys)
  - Qualtrics privacy policy: https://www.qualtrics.com/privacy-statement/
- Twilio (for text messages)
  - o Twilio privacy policy: <a href="https://www.twilio.com/legal/archive/2018-05-14/privacy">https://www.twilio.com/legal/archive/2018-05-14/privacy</a>

By signing this consent form you are allowing the study team to provide the vendors with your contact information to mail you something to your address, email you, or text you. Not all of these companies have signed a confidentiality agreement with us. However, they each have their own privacy statements. They will not know the results of any of your tests or other research information.

We are also asking you to use the MyFitnessPal website, which will require you to create a free account using your email address. You'll be asked to use MyFitnessPal throughout the program even if you didn't use it to track your food during the enrollment steps.

# How will your blood samples be stored and used?

Your blood will be frozen and stored until it is sent to a lab for testing. Blood tests may include (1) liver function tests (2) diabetes related tests and (3) cholesterol related tests. Additional blood will be drawn to assess effects on an appetite suppressing hormone. Also, blood will be drawn for induced pluripotent stem (iPS) cell tests, as well, if you agree to participate in this component of our research.

# Will I receive my test results?

All blood test and MRI results will be posted to your patient portal through Michigan Medicine. You will not receive the results of the iPS cell or hormone testing, as these are experimental.

# What are my responsibilities?

As a subject participating in this research study, you have certain responsibilities, such as ensuring that you arrive at all of your scheduled appointments, follow the study meal plans, and report any side effects you may experience to the study team during the study.

# 4.2 How much of my time will be needed to take part in this study?

Your participation in the study will take about 6 months. You will have up to two baseline and up to two post-study visits, each lasting 1-2 hours, and the 4-month diet and lifestyle program. Participation in the diet and lifestyle program will take varying amounts of time, but the class materials may take 1-2 hours to read and apply each week.

If you would like to participate in the exit interview after the study is completed, we will set up a time for a phone call with a study team member. The interview will be audio recorded; if you decline to be recorded, we will not proceed with the interview. The interview will take approximately 30 minutes to complete. The recording of the interview will be sent to a transcription company who will send us the finished transcriptions and then all audio files will be deleted. We will avoid using any identifiable information in the interview.

# 4.3 When will my participation in the study be over?

The study period is about 6 months in duration. Your participation in the study will end at this time.

# 4.4 What will happen with my information and/or biospecimens used in this study?

Your biospecimens and collected information may be shared with the Michigan Nutrition Obesity Research Center or the National Institutes of Health, who sponsor this study.

Most of your blood will be destroyed at the end of the study. However, if you agree to participate in iPS cell testing, some of your blood may be kept in Dr. Speliotes' lab indefinitely. Dr. Speliotes is an investigator on this study. Cells multiply by dividing in two, and the genetic material is replicated every time a cell divides. It is possible that iPS cell lines, which can live indefinitely, may contain all or part of your DNA. You should be aware that your tissues, cells or other materials derived from these tissues may be kept for many years.

In most cases, your tissue or cells will be stored indefinitely in Dr. Speliotes' laboratory, located at the University of Michigan Medical School. Only Dr. Speliotes and her study staff will know your identity. After your blood is brought to the lab, your identifying information will be removed and will be labeled with a code instead.

With appropriate permissions, your biospecimens and collected information may also be shared with other researchers, here, around the world, and with companies.

Your identifiable private information or identifiable biospecimens, iPS cells included, may be stripped of identifiers and used for future research studies or distributed to another researcher for future research studies without additional informed consent.

Your stored tissues and cells and the iPS cell lines derived from them could be used in future related and unrelated studies, which are not foreseeable now. There are several possible research uses for tissues and cells donated for pluripotent stem cell research, including:

- Injecting or transplanting the stem cells into animals for research-only purposes.
- Testing for genetic and DNA composition. Genes may be analyzed and/or manipulated to study normal function or development.
- Patenting derived stem cells, which contain your DNA, for scientific or medical use.
  - If any new products, tests, discoveries or patents that result from this research have potential commercial value, you will not share in any financial benefits. You will not receive patent rights. You will not have control over the product sales and uses (except as stated in this consent).
- Creating a tissue-specific stem cell line, which could be transplanted into another human for the purpose of treating people with NAFLD or other disorders.
- Other, currently unknown uses. Science is always evolving and it is therefore difficult to determine exactly how these cells will be used in the future.

# 5. INFORMATION ABOUT STUDY RISKS AND BENEFITS

# 5.1 What risks will I face by taking part in the study? What will the researchers do to protect me against these risks?

- 1. <u>Blood draw:</u> Your blood draw is considered standard of care for NAFLD. It includes a possibility of bleeding, bruising, and dizziness. It is common for the site of the test to bleed after the blood sample has been taken; however, this should stop fairly quickly after a cotton wool pad or gauze patch has been placed on the wound. Mild bruising around the area where the needle went into the vein and/or slight dizziness during or after a blood test is fairly common. If you are feeling faint before or during a blood test, tell the person taking your blood so that they can help you.
- 2. <u>Liver MRI:</u> If you have implanted metal objects such as a pacemaker, artificial limbs, or metal joints, you will not be able to have an MRI done, and will not be able to take part in this research. The MRIs for this study do not include any contrast (injected dye) and are completely non-invasive. Common risks of MRI include: feeling fearful of being in a small enclosed space (claustrophobia) when you are lying inside the MRI scanner, feeling uncomfortable because of the loud noises made by the machines, and feeling uncomfortable with the physical sensations you may feel during the process. Some people may feel claustrophobic or may not be able to hold their breath during image capture. The MRI technician will provide you with blankets to

make you feel as comfortable as possible. You will be able to talk to the technician and can let them know right away if you feel you need to stop and get out of the scanner. You will also wear earplugs and headphones to reduce the loud noises made by the scanner. Sometimes, subjects report a temporary, slight dizziness, light-headedness or nausea during or immediately after the scanning session. If you feel dizzy or light-headed, the MRI technician will help you get up slowly from the scanner. You won't feel the magnetic field or radio waves. Most MRI machines consist of a large magnet shaped like a tunnel. You lie on a table that slides into the tunnel. A computer creates a composite, three-dimensional representation of your body. Two-dimensional images are then created and displayed on a monitor and/or converted into photographic film for further viewing and analysis. If you feel uncomfortable, please let the technician know, so that they can adjust or stop the scan. The MRI technician will also review the procedure with you in-depth. The scan should take no more than an hour, but plan for a 2 hour appointment.

- 3. <u>Questionnaires:</u> Some of the questions may make you uncomfortable or upset, but you are free to decline to answer any questions you do not wish to answer or to discontinue your participation at any time.
- 4. <u>Diet:</u> As you change your diet you may experience some side effects such as constipation, headache, bad breath, and muscle cramps. These symptoms usually go away after the first couple weeks. If this happens, you can talk to the study staff. Additionally, kidney stones are common in the general population you are advised to follow diet recommendations, eat a normal amount of protein, and increase your water intake to avoid kidney stones during the study. Recommendations for daily water intake will be included in the lesson for week 2. The study staff will provide resources for eating a healthful, very low-carbohydrate diet and aid in management of any side effects, though you can and should consult your doctor if any side effects are concerning to you or become severe.
- 5. <u>Dietary changes:</u> You could find it difficult to change your diet. Also, your friends or family may not support the changes you are making to your diet or lifestyle. If this happens, you can speak to study staff about this.
- Home assignments: You may find it inconvenient to complete the home assignments. Also, you could experience distressing emotions during some of the home assignments. If this happens, you can stop and speak to the study staff.
- 7. <u>Audio recording:</u> If you participate in the exit interview, your interview will be recorded. This recording will be saved on encrypted, University computers, sent to an external transcription company, and then deleted. We will avoid using any personal information in the interview and if names are used, they will not be included in the transcript. Recording and transcription comes with the possibility of loss of privacy, though this is rare.

As with any research study, there may be additional risks that are unknown or unexpected.

Additionally, there may be a risk of loss to confidentiality or privacy. See Section 9 of this document for more information on how the study team will protect your confidentiality and privacy.

5.2 What happens if I get hurt, become sick, or have other problems as a result of this research?

The researchers have taken steps to minimize the risks of this study. You may still have problems or side effects, even when the researchers are careful to avoid them. Please tell the researchers listed in Section 10 about any injuries, side effects, or other problems that you have during this study. You should also tell your regular doctors.

We will ask you measure your ketone levels (with a urine strip) and your body weight (with a scale we send you) in order to assess how your body changes in response to the diet and lifestyle recommendations. If you're taking glucose-lowering medications other than metformin, we'll send you a blood-glucose monitor so you can keep track of your blood glucose and adjust your medication with the help of your primary care physician, if necessary. You'll report your highest and lowest blood glucose readings while fasting and 2 hours after eating each week. If you are taking TZDs, DPP4 inhibitors, GLP-1 agonists, you will continue your medications as normal and track your blood glucose throughout the trial. If you are taking other glucose-lowering medications, such as sulfonylureas, meglitinides, and SGLT-2 inhibitors, you'll be advised to stop those medications to ensure your blood sugar doesn't get too low as you switch your diet. A study physician, Dr. Dina Hafez Griauzde, will work with you if your blood sugar appears too high or low throughout the study and your doctor will be informed of your medication adjustments. We will encourage you to reach out to your primary care physician if any of these changes appear to negatively impact your overall health or if you experience persistent or severe side effects. You'll keep anything that we send you at the end of the study (including the scale and glucose monitor).

# 5.3 If I take part in this study, can I also participate in other studies?

<u>Being in more than one research study at the same time, or even at different times, may increase the risks to you. It may also affect the results of the studies</u>. You should not take part in more than one study without approval from the researchers involved in each study.

### 5.4 How could I benefit if I take part in this study? How could others benefit?

You may not receive any personal benefits from being in this study. However, others may benefit from the knowledge gained from this study.

Many participants may receive benefits from their participation in this study. These may include reduced blood pressure, improved glycemic (sugar) control, weight loss, reduced risk for diabetes complications, and decreased feelings of stress, but this cannot be guaranteed. The information that you provide may also provide benefit to other individuals like you, by helping health professionals and researchers better understand how to help people with these conditions improve their health and lower their risk for complications.

# 5.5 Will the researchers tell me if they learn of new information that could change my willingness to stay in this study?

Yes, the researchers will tell you if they learn of important new information that may change your willingness to stay in this study. If new information is provided to you after you have joined the study, it is possible that you may be asked to sign a new consent form that includes the new information.

# 6. ALTERNATIVES TO PARTICIPATING IN THE STUDY

#### 6.1 If I decide not to take part in this study, what other options do I have?

You are free to choose not to participate in this study. If you decide not to take part in this study, there will be no penalty to you. You will not lose any of your regular benefits, and you can still get care the way you usually do.

There may be other ways of treating your condition. These include talking to your primary care physician about your non-alcoholic fatty liver disease. Although the WELL program is available as part of this clinical study, you should check with the researcher and/or your primary care physician to discuss your options including how to obtain any alternative treatments and whether they must be obtained through a physician or require medical supervision.

### 7. ENDING THE STUDY

# 7.1 If I want to stop participating in the study, what should I do?

You are free to leave the study at any time. If you leave the study before it is finished, there will be no penalty to you. You will not lose any benefits to which you may otherwise be entitled. If you choose to tell the researchers why you are leaving the study, your reasons for leaving may be kept as part of the study record. If you decide to leave the study before it is finished, please tell one of the persons listed in Section 10 "Contact Information".

# 7.2 Could there be any harm to me if I decide to leave the study before it is finished?

No harm will come to you if you decide to leave the study before it is finished. We may ask you why you've decided to stop your participation in order to better understand how we could improve the program for future participants.

# 7.3 Could the researchers take me out of the study even if I want to continue to participate?

Yes. There are many reasons why the researchers may need to end your participation in the study. Some examples are:

- The researcher believes that it is not in your best interest to stay in the study.
- You become ineligible to participate.
- Your condition changes and you need treatment that is not allowed while you are taking part in the study.
- You do not follow instructions from the researchers.
- The study is suspended or canceled.

# 8. FINANCIAL INFORMATION

# 8.1 Who will pay for the costs of the study? Will I or my health plan be billed for any costs of the study?

The medical care that you receive in this study is a part of your standard of care. You or your health plan will be responsible for all the things you would have paid for even if you were not in the study, like:

- The 2 office visits, your first MRI, and fasting blood tests (liver function tests, diabetes related tests and cholesterol related tests).
- Any visits to your personal physician if there are changes that negatively impact your overall health while you are on the study.

The research will pay for your second MRI, both insulin tests, and the extra blood drawn for research.

If you get a bill that you think is incorrect, please contact the research team.

Health care given during the study as part of your regular care. You are your health plan will also be responsible for:

Items or services needed to give you study drugs or devices

IRBMED Informed Consent Template—3-9-2018
Instructions revised 3-9-2018
DO NOT CHANGE THIS FIELD—IRB USE ONLY

- Monitoring for side effects or other problems
- Deductibles or co-pays for these items or services

If you do not have a health plan, or if you think your health plan may not cover these costs during the study, please talk to the researchers listed in Section 10 below or call your health plan's medical reviewer.

By signing this form, you do not give up your right to seek payment if you are harmed as a result of being in this study.

# 8.2 Will I be paid or given anything for taking part in this study?

If you complete your screening eligibility tasks and you are ineligible after your second appointment, you will be paid \$20 in an Amazon gift card.

After the 4-month study is completed and you complete **all** final tasks, you will receive \$100. You will be paid with an Amazon.com gift certificate that will be emailed to you. In addition, you will be able to keep any materials that you may receive as part of the study, including the blood glucose monitor, if applicable.

If you withdraw early from the study for any reason or you do not complete the 4-month tasks, you will not receive any compensation. You will be able to keep any materials you have received as part of the study.

# 8.3 Who could profit or financially benefit from the study results?

Dr. Laura Saslow's partner, Mr. Hovig Bayandorian, is an inventor of software being used in this research and provides this study a services agreement.

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the use of the data or discoveries. You will not have rights to these discoveries or any proceeds from them.

# 9. CONFIDENTIALITY OF SUBJECT RECORDS AND AUTHORIZATION TO RELEASE YOUR PROTECTED HEALTH INFORMATION

The information below describes how the confidentiality of your research records will be protected in this study, and any sub-studies described in this document.

# 9.1 How will the researchers protect my information?

Your research information will be kept in a locked filing cabinets or stored on encrypted servers and computers accessible only by study staff. Information from your medical exam, blood tests, and MRI will become part of your regular medical record. You will receive a participant ID that will be used in place of your name on study related communications. All information is protected and confidential.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or

local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by Michigan Nutrition Obesity Research Center (the sponsor), which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law.

The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document.

Your information will be stored on encrypted servers and computers accessible only by study staff. We will mail class information weekly using email and may send you text messages and you may email or call us about questions pertaining to the study or your health. Participation in research may involve a loss of privacy, but information about you will be handled as confidentially as possible.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov/">http://www.clinicaltrials.gov/</a>, as required by U.S. Law. This web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this website at any time.

# 9.2 What protected health information (PHI) about me could be seen by the researchers or by other people? Why? Who might see it?

Signing this form gives the researchers your permission to obtain, use, and share information about you for this study, and is required in order for you to take part in the study.

Medical information and billing records are protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA). This type of information is called protected health information (PHI). PHI about you may be obtained from any hospital, doctor, and other health care provider involved in your care, including:

- Hospital/doctor's office records, including test results (X-rays, blood tests, urine tests, etc.)
- Health plan/health insurance records
- All records relating to your condition, the treatment you have received, and your response to the treatment
- Billing information
- Demographic information
- Personal identifiers

There are many reasons why information about you may be used or seen by the researchers or others during or after this study. Examples include:

- The researchers may need the information to make sure you can take part in the study.
- The researchers may need the information to check your test results or look for side effects.
- University, Food and Drug Administration (FDA) and/or other government officials, auditors, and/or the IRB may need the information to make sure that the study is done in a safe and proper manner.
- Study sponsors or funders, or safety monitors or committees, may need the information to:
  - Make sure the study is done safely and properly
  - Learn more about side effects
  - Analyze the results of the study
- Insurance companies or other organizations may need the information in order to pay your medical bills or other costs of your participation in the study.
- The researchers may need to use the information to create a databank of information about your condition or its treatment.
- Information about your study participation may be included in your regular UMHS medical record
- If you receive any payments for taking part in this study, the University of Michigan accounting department may need your name, address, Social Security number, payment amount, and related information for tax reporting purposes.
- Federal or State law may require the study team to give information to government agencies. For example, to prevent harm to you or others, or for public health reasons.
- As mentioned above, some of your study materials and emails will be sent directly to you through vendors such as Amazon and Zinc.io (for mailing gift certificates and cookbooks, as well as for encrypted storage), BodyTrace (body weight scale), GSuite/Gmail and Postmarkapp (for emails), Qualtrics (for surveys), and Twilio (for text messages). By signing this consent form you are allowing the study team to provide the vendors with your contact information as needed to mail something to your physical address, email you, or text you.

Additionally, because the appointments you'll be attending in this study are part of your standard of care, the information about these appointments, including any potential diagnoses and the results of your blood tests and MRIs will become part of your medical record.

The results of this study could be published in an article, but would not include any information that would let others know who you are.

# 9.3 What happens to information about me after the study is over or if I cancel my permission to use my PHI?

As a rule, the researchers will not continue to use or disclose information about you, but will keep it secure until it is destroyed. Sometimes, it may be necessary for information about you to continue to be used or disclosed, even after you have canceled your permission or the study is over.

Examples of reasons for this include:

- To avoid losing study results that have already included your information.
- To provide limited information for research, education, or other activities. (This information
  would not include your name, social security number, or anything else that could let others
  know who you are.)

• To help University and government officials make sure that the study was conducted properly. As long as your information is kept within the University of Michigan Health System, it is protected by the Health System's privacy policies. For more information about these policies, ask for a copy of the University of Michigan "Notice of Privacy Practices". This information is also available on the web at <a href="http://www.uofmhealth.org/patient+and+visitor+guide/hipaa">http://www.uofmhealth.org/patient+and+visitor+guide/hipaa</a>. Note that once your information has been shared with others as described under Question 9.2, it may no longer be protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA).

# 9.4 When does my permission to use my PHI expire?

Your permission expires at the end of the study, unless you cancel it sooner. You may cancel your permission at any time by writing to the researchers listed in Section 10 "Contact Information" (below). If you withdraw your permission, you may no longer be eligible to participate in this study.

### **10. CONTACT INFORMATION**

# 10.1 Who can I contact about this study?

Please contact the researchers listed below to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Talk about study-related costs to you or your health plan
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

# Principal Investigator:

Laura Saslow; Mailing Address: Office 2178, 400 N Ingalls St, Ann Arbor, MI, 48109;
 Telephone: 734-764-7836

Study Coordinator:

• Jamie Krinock

Telephone: 734-763-4571

# You may also express a question or concern about a study by contacting the Institutional Review Board listed below:

University of Michigan Medical School Institutional Review Board (IRBMED)

2800 Plymouth Road Building 520, Room 3214 Ann Arbor, MI 48109-2800

Telephone: 734-763-4768 (For International Studies, include the appropriate calling codes.)

Fax: 734-763-1234

email: <a href="mailto:irbmed@umich.edu">irbmed@umich.edu</a>

If you are concerned about a possible violation of your privacy or concerned about a study you may contact the University of Michigan Health System Compliance Help Line at 1-866-990-0111. When you call or write about a concern, please provide as much information as possible, including the name of the researcher, the IRBMED number (at the top of this form), and details about the problem. This will help University officials to look into your concern. When reporting a concern, you do not have to give your name unless you want to.

# 11. RECORD OF INFORMATION PROVIDED

# 11.1 What documents will be given to me?

Your signature in the next section means that you have received copies of all of the following documents:

This "Consent to be Part of a Research Study" document. (*Note: In addition to the copy you receive, copies of this document will be stored in a separate confidential research file and may be entered into your regular University of Michigan medical record.*) You will have this document as a downloadable pdf file.

12. SIGNATURES

| Sig-A |
|---|
| Consent to Participate in the Research Study |
| I understand the information printed on this form. I have discussed this study, its risks and potential benefits, and my other choices with [NAME OF STUDY TEAM MEMBER OBTAINING CONSENT] My questions so far have been answered. I understand that if I have more questions or concerns about the study or my participation as a research subject, I may contact one of the people listed in Section 10 (above). I understand that I will receive a copy of this form at the time I sign it and later upon request. I understand that if my ability to consent or assent for myself changes, either I or my legal representative may be asked to reconsent prior to my continued participation in this study. Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |
| Sig-B |
| Consent to audio recording solely for purposes of this research This study involves optional audio recording. If you do not agree to be recorded, you CAN STILL take part in the study, but you will not be able to participate in the optional exit interview. You can opt out of the interview later, if you change your mind. |
| Yes, I agree to audio recorded. |
| No, I do not agree to be audio recorded. |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |

IRBMED Informed Consent Template—3-9-2018

Instructions revised 3-9-2018

DO NOT CHANGE THIS FIELD—IRB USE ONLY

| Sig-C |
|---|
| Consent for Participating in an Optional Induced Pluripotent Stem (iPS) Cell Research This project involves optional participation in iPS cell research. I understand that it is my choice whether or not to take part in this study activity. I understand that if my ability to consent for myself changes, I may be asked to re-consent prior to my continued participation in this study. |
| Yes, I agree to take part in the optional iPS cell research. |
| No, I do not agree to take part in the optional iPS cell research. |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |
| Sig-G<br>Principal Investigator or Designee |
| I have provided this participant and/or his/her legally authorized representative(s) with information about this study that I believe to be accurate and complete. The participant and/or his/her legally authorized representative(s) indicated that he or she understands the nature of the study, including risks and benefits of participating. |
| Printed Legal Name: |
| Title: |
| Signature: |
| Date of Signature (mm/dd/yy): |